CLINICAL TRIAL: NCT05619068
Title: Imaging Investigation on the Evolution and Prognosis of Moyamoya Disease
Brief Title: The Evolution and Prognosis of Moyamoya Disease
Status: Recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Xin Lou, Chairman, Chinese PLA General Hospital
Other Study IDs: MMD-301
Record Dates: First submitted 2022-11-05; First posted 2022-11-16 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Moyamoya Disease; Revascularization; Cognitive Impairment; Functional Impairment
Keywords: Moyamoya disease; Revascularization; Cognitive impairment; Functional impairment
MeSH Terms: conditions — Moyamoya Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Medical treatment group: Conservative medical treatment
- Surgical treatment group: Direct revascularization, indirect revascularization or combined revascularization

SUMMARY:
To investigate the evolution of imaging appearances and cognitive function of Moyamoya disease (MMD) and to establish a prognosis evaluation system based on imaging biomarkers in MMD. The study may be helpful to optimize and improve the diagnosis and pretreatment assessment of MMD, and provide an important theoretical supplement to the existing guidelines for the management of MMD.

DETAILED DESCRIPTION:
Moyamoya disease (MMD) is a chronic progressive cerebrovascular disease of unknown etiology. It is characterized by chronic progressive stenosis or occlusion of bilateral internal carotid arteries and abnormal puff vessels at the base of the brain. MMD is one of the important causes of cerebrovascular accident in young and middle-aged people, which leads to about 22% of stroke. With the development of neurosurgery, revascularization can effectively reduce the risk of stroke and other cerebrovascular accidents by increasing cerebral perfusion. Therefore, this project is expected to improve the diagnosis and pretreatment assessment of MMD from the traditional level of symptomatology to the level of brain cognitive function through new imaging methods and clinical approaches. The study of cognitive function changes in follow-up period or after revascularization, which is of great scientific significance for understanding the plasticity of cognitive function under different cerebral perfusion conditions, will also be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Patients with MMD: Conventional angiography or MRI examination conforms to the Guidelines for Diagnosis and Treatment of MMD (Neurol Med Chir (Tokyo) 52, 245-266, 2012), It is characterized by stenosis or occlusion of the end of the internal carotid artery, anterior cerebral artery and/or the beginning of the middle cerebral artery of unknown cause, accompanied by dilatation of the perforating artery at the base of the brain or of capillaries on the surface of the brain, i.e., the formation of smoke vessels. Sign the informed consent. Older than 10 and younger than 60. The education level of patients reached primary school or above (years of education ≥6).

Exclusion Criteria:

* Patients with massive cerebral infarction, multiple paraventricular ischemic foci, or significantly enlarged ventricular hydrocephalus after intracerebral hemorrhage. Patients with vascular diseases caused by immune system disease. Patients can not cooperate to complete the cognitive function test. There are other neuropsychiatric diseases that affect cognitive function (such as Alzheimer's disease, Parkinson's disease, depression, anxiety disorder, cerebral hemorrhage, hydrocephalus, craniocerebral trauma, etc.). Patients with contraindications of magnetic resonance examination (patients with pacemakers, nerve stimulators, artificial metal heart valves and other metal foreign bodies) or unable to complete image collection.

Ages: 10 Years to 60 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients confirmed with Moyamoya disease.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Cognitive decline | 1-5 years
  Cognitive decline was defined as decreasing in any of the scale below. Choice reaction time was used as the baseline condition and the index of movement ability. Nonverbal matrix reasoning was used to assess general intelligence and reasoning ability. The Eight-item Interview to Differentiate Aging and Dementia questionnaire was used to determine the degree of cognitive decline in daily life. The mental rotation was used to evaluate the visual-spatial ability. Verbal working memory was used to measure working memory capacity. All cognitive assessment were tested using an Online Psychological Experimental System.

SECONDARY OUTCOMES:
Changes of functional connectivity | 1-5 years
  Changes of the pattern of functional connectivity assessed by functional magnetic resonance imaging from baseline to the follow-up scan.
Changes of perfusion status | 1-5 years
  Changes of the severity of hypoperfusion (hypoperfusion volume) on magnetic resonance imaging from baseline to the follow-up scan.

CONTACTS AND LOCATIONS:
Overall Officials: Lou Xin, MD, PhD, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China